CLINICAL TRIAL: NCT03630926
Title: Evaluation of the NV-VPAC1 Prostate Cancer (PCa) Urine Diagnostic Test in Subjects With Biopsy-confirmed Prostate Cancer, Benign Prostatic Hypertrophy, or Bladder/Kidney Stones
Acronym: VPAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: NuView Diagnostics (Unknown)
Responsible Party: Principal Investigator, JAY BISHOFF, Director of Intermountain Urological Institute, Intermountain Health Care, Inc.
Other Study IDs: VPAC
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer; Benign Prostatic Hypertrophy; Bladder Stones; Kidney Stones
Keywords: NV-VPAC1 Prostate Cancer Urine Diagnostic test
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia; Urinary Bladder Calculi; Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prostate Cancer (PCa): Comprised of men with biopsy-confirmed PCa who are scheduled for prostatectomy.
  Interventions: Diagnostic Test: NV-VPAC1 PCa Urine Diagnostic Test
- Benign Prostatic Hypertrophy (BPH): comprosed of men with benign prostatic hypertrophy (BPH) who are scheduled for transurethral resection of the prostate (TURP).
  Interventions: Diagnostic Test: NV-VPAC1 PCa Urine Diagnostic Test
- Bladder/kidney stone: Comprised of men or women with bladder/kidney stones who are scheduled for a cystoscopy.
  Interventions: Diagnostic Test: NV-VPAC1 PCa Urine Diagnostic Test

INTERVENTIONS:
Diagnostic Test: NV-VPAC1 PCa Urine Diagnostic Test — The NV-VPAC1 PCa Urine Diagnostic Test is intended for use by clinicians to detect the presence of prostate cancer cells shed in voided urine of men at risk for prostate cancer.

SUMMARY:
This is a double-blind, study to evaluate the performance of NV-VPAC1 PCa Urine Diagnostic Test in three distinct populations being treated at the Intermountain Urology Clinic. The first population (positive control) is comprised of men with biopsy-confirmed PCa who are scheduled for prostatectomy. The second population (negative control) is comprised of men with benign prostatic hypertrophy (BPH) who are scheduled for transurethral resection of the prostate (TURP). The third population (negative control) is comprised of men or women with bladder/kidney stones who are scheduled for a cystoscopy.

ELIGIBILITY:
Subjects with prostate cancer

Inclusion Criteria:

* Males 18-80 years of age
* Biopsy-confirmed prostate cancer
* Scheduled within 2 weeks for prostatectomy
* Signed informed consent

Exclusion Criteria:

* Presence or history of another cancer diagnosis, with the exception of certain skin cancers
* Currently treated with finasteride (Proscar®, Propecia®), dutasteride (Avodart®) or anti-androgen therapy (Lupron®)
* Participated in a clinical study with an investigational drug within 2 weeks of the screening visit.

Subjects with benign prostatic hypertrophy

Inclusion Criteria:

* Males 18-80 years of age
* Diagnosis of BPH made by clinical symptoms (e.g., enlarged prostate, dribbling urine stream, frequent and urgent urination)
* Scheduled within 2 weeks for TURP
* Signed informed consent

Exclusion Criteria:

* Presence or history of any cancer diagnosis, with the exception of certain skin cancers
* Currently treated with finasteride (Proscar®, Propecia®) or dutasteride (Avodart®)
* Participated in a clinical study with an investigational drug within 2 weeks of the screening visit.

Subjects with bladder/kidney stones

Inclusion Criteria:

* Males or females 18-80 years of age
* Diagnosed with bladder/kidney stones
* Scheduled within 2 weeks for cystoscopy
* Signed informed consent

Exclusion Criteria:

* Presence or history of any cancer diagnosis, with the exception of certain skin cancers
* Participated in a clinical study with an investigational drug within 2 weeks of the screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy-confirmed prostate cancer, patients with BPH, and patients with bladder/kidney stones
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Degree of association of the presence of orange fluorescent positive cells shed in voided urine and lack of association of orange fluorescent positive cells in men diagnosed with BPH or in individuals with bladder/kidney stones | 6 months
  Degree of association of the presence of orange fluorescent positive cells shed in voided urine of men with biopsy-proven PCa and lack of association of orange fluorescent positive cells in men diagnosed with BPH or in individuals with bladder/kidney stones

SECONDARY OUTCOMES:
Association between PSA levels and NV-VPAC1 test results. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jay Bishoff, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States